CLINICAL TRIAL: NCT05876026
Title: MRI T1 Relaxation Times in Evaluating Neoadjuvant Treatment of Rectal Cancer
Brief Title: MRI T1 Relaxation Time in Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: T1 relaxation MRI
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Rectal Cancer; Locally Advanced Rectal Carcinoma
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the T1 relaxation time and T1 relaxation time properties of the disease in people with locally advanced rectal cancer. The main question it aims to answer is:

Does MRI T1 relaxation time have a high diagnostic performance in recognizing fibrosis as a complete response to neoadjuvant treatment of rectal cancer?

Participants will receive standard neoadjuvant treatment and be part of the standard examination programme regarding rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* rectal cancer, age >18 years

Exclusion Criteria:

* contraindications for MRI (pacemaker, claustrophobia, implanted medical injectors and nerve stimulators),
* previous radiochemotherapy or another disease which investigator judges inappropriate for the persons continued participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with rectal cancer (>18 years of age) and no previous history of radiochemotherapy. The population will consist of people from the Region of Southern Denmark.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Difference in T1 relaxation time (ms) in the rectal cancer tumor measured in IntelliSpace-software before and after neoadjuvant radiochemotherapy. | 6 to 8 weeks.
  An MRI T1 relaxation time-map is performed on each participant. The data is transferred to IntelliSpace-software for measurement and mapping. It is measured in miliseconds (ms) before and after neoadjuvant treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Søren Rafaelsen, DMSc, Study Chair — Vejle Hospital
Locations (1):
- Vejle Hospital, Vejle, Jylland, Denmark